CLINICAL TRIAL: NCT01965340
Title: Impact of Therapeutic Drug Monitoring on Anti-Infective Agents Amongst Severely Burned Patients Requiring ICU Admission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Anne Fournier, Anne Fournier, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 195/13
Record Dates: First submitted 2013-09-27; First posted 2013-10-18 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Burn
Keywords: patients
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with systematic TDM of anti-infective agents (Experimental): Patients with systematic TDM of anti-infective agents and dosages adapted accordingly
  Interventions: Other: Systematic Therapeutic Drug Monitoring for the intervention group
- Patients treated as usual (No Intervention)

INTERVENTIONS:
Other: Systematic Therapeutic Drug Monitoring for the intervention group
  Arms: Patients with systematic TDM of anti-infective agents

SUMMARY:
Sepsis is the major cause of morbidity and mortality amongst burn patients. Burn shock and respiratory failure that used to be the major cause of mortality have progressively been replaced by sepsis and multiple organ failure. It is not rare that treatment failures occurs several weeks, or even months after injury as a consequence of sepsis usually caused by multi-drug resistant (MDR) microorganisms. Introduction of early surgery combined with topical and systemic antibiotherapy dramatically enhanced survival from sepsis after burn trauma, but further improvement is impaired by the rapid development of hard-to-treat MDR bacteria.

Correct prescription of anti-infective agents could be one way to curb the steadily increasing development of multidrug resistance. Administration of antibiotic to burn patient is complex: they frequently suffer from kidney dysfunction, they usually experience tremendous shifts of liquids between intra-vascular - inter-cellular and intra-cellular compartments, they often are hypo-albumin and protein-emic, and finally they present with a profoundly modified metabolism. All those aspects make this particular population of patients at high risk of both under or over prescription.

Monitoring of drug concentrations in the plasma of patients, so-called TDM for Therapeutic Drug Monitoring, has been introduced to clinical practice for several decades primarily to avoid toxicity of a small number of drugs with narrow therapeutic windows. However, with the increasing availability of detection techniques, the number of drugs that can be measured in the plasma of patients has grown tremendously over the last decade. As a consequence, it is currently possible to monitor drug concentrations not only to prevent toxicity, but also to improve efficacy. For instance, several studies demonstrated that TDM improved antibiotic prescription in different populations of hospitalized patients, including critically ill patients, with a direct impact on outcome.

Such studies amongst burn patients are however lacking, although this particular population is at high risk to suffer from mis-prescription. We thus hypothesize that systematic TDM could improve antibiotic prescription in this peculiar population. To this end, we propose to implement a 3-year prospective, randomized, mono-centric, clinical trial that will analyze the impact of systematic TDM on anti-infective agent prescription amongst burned patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult burn patients (≥ 18 years) admitted to the University Hospital of Lausanne during the study period receiving systemic anti-infectives agents for which TDM is available will be included.

Exclusion Criteria:

* Patients not receiving systemic anti-infective agents therapy
* Patients with length of hospital stay <72 hours
* Patients refusing to give their written consent (or for which the therapeutic representative refuses) or incapable of understanding and lack of legal representative
* Pregnant or breastfeeding women
* Children <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Time required to achieve anti-infective plasma concentrations in the target | Up to 3 years
Numbers of concentrations within the target during an anti-infective agents course | Up to 3 years

SECONDARY OUTCOMES:
Anti-infective agents consumption | Up to 3 years
Development of antibiotic resistance | Up to 3 years
Length of ICU stay based on TBSA | Up to 3 years
Characterization of the pharmacokinetic profile of most widely used antibiotics | Up to 3 years
Concentration - efficacy analysis | Up to 3 years
  Population pharmacokinetic (NONMEM software)
Failure / resolution rate of infectious episodes | Up to 3 years
Concentration - toxicity analysis | Up to 3 years
  Population pharmacokinetic (NONMEM software)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Fournier A, Goutelle S, Que YA, Eggimann P, Pantet O, Sadeghipour F, Voirol P, Csajka C. Population Pharmacokinetic Study of Amoxicillin-Treated Burn Patients Hospitalized at a Swiss Tertiary-Care Center. Antimicrob Agents Chemother. 2018 Aug 27;62(9):e00505-18. doi: 10.1128/AAC.00505-18. Print 2018 Sep. PMID 29914948
- [Derived] Fournier A, Eggimann P, Pantet O, Pagani JL, Dupuis-Lozeron E, Pannatier A, Sadeghipour F, Voirol P, Que YA. Impact of Real-Time Therapeutic Drug Monitoring on the Prescription of Antibiotics in Burn Patients Requiring Admission to the Intensive Care Unit. Antimicrob Agents Chemother. 2018 Feb 23;62(3):e01818-17. doi: 10.1128/AAC.01818-17. Print 2018 Mar. PMID 29263079